CLINICAL TRIAL: NCT06422104
Title: Development of Mechanistically Informed Therapy for Task-Specific Dystonia Using Noninvasive Neuromodulation
Brief Title: Neuromodulation Therapy for Task-Specific Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Dystonia Coalition (Other); Dystonia Study Group (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00094131
Record Dates: First submitted 2024-04-24; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Isolated Focal Hand Dystonia
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind cross-over design with participants receiving TMS at two cortical locations.
Who Masked: Participant, Outcomes Assessor
Masking Description: The TMS intensity and cortical location delivered at each TMS visit will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- 10 Hz rTMS to premotor cortex (Active Comparator): 10 Hz rTMS to premotor cortex
  Interventions: Device: Repetitive transcranial magnetic stimulation
- 10 Hz rTMS to primary somatosensory cortex (Active Comparator): 10 Hz rTMS to primary somatosensory cortex
  Interventions: Device: Repetitive transcranial magnetic stimulation
- 0.7 Hz rTMS to premotor cortex (Active Comparator): 0.7 Hz rTMS to premotor cortex
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — 10 Hz repetitive TMS will be delivered for 20 minutes per session and 0.7 Hz for 20 minutes per session

SUMMARY:
This study aims to apply a non-invasive brain stimulation technology called repetitive Transcranial Magnetic Stimulation (rTMS) in patients with focal hand dystonia (FHD). The goal of the study is to identify which cortical target (premotor cortex (PMC) or primary somatosensory cortex (PSC)) will show benefit after active rTMS compared to sham rTMS. A secondary goal of the study is to understand if 10 Hz rTMS can show behavioral benefit compared to sham rTMS. The study will evaluate rTMS response using measures if writing on a sensor tablet, examiner and patient dystonia rating scales and brain imaging scan (functional MRI) to understand brain changes after rTMS. Safety measures include adherence to TMS guidelines and thorough medical screening to prevent seizures.

DETAILED DESCRIPTION:
The primary objective of this study is to develop rTMS for FHD. The focus is to assess whether stimulating the PMC or PSC will show greater improvement in writing behavior. This research builds upon prior studies that have demonstrated improvement in behavior after rTMS to PMC and PSC. The study includes five sequential visits:

* Visit 1 behavior writing measures and dystonia rating scales.
* Visit 2 includes task-based functional MRI brain scans to develop cortical target for rTMS sessions.
* Visits 3, 4, and 5: FHD participants receive 10 Hz rTMS to PMC, PSC and sham rTMS to PMC in a cross over design with at minimum one week of washout between sessions. Participants complete behavior writing measures and rating scales on same day before and after each TMS session and an fMRI after each TMS session. Up to 5 Healthy Volunteers were recruited to help develop the TMS visits.

The information in this record reflects Visits 2-5

ELIGIBILITY:
Inclusion Criteria:

* Healthy Control Participants:

  1. 18yrs and older
  2. Left or Right hand dominance
  3. Age-matched to Focal Hand dystonia patients
  4. Must be able to sign informed consent
  5. Must be literate
* Focal Hand dystonia Patients:

  1. 18yrs and older
  2. Left or Right hand dominance
  3. Diagnosed with Writer's Cramp dystonia in left or right hand
  4. Must be able to sign informed consent
  5. Must be literate

Exclusion Criteria:

Healthy Control Participants (visits 2, 3, 4, and 5) and Focal Hand dystonia Patients (visits 2, 3, 4, and 5):

1. Other neurological movement disorders diagnoses including other types of dystonia, Parkinsonism, or essential tremor
2. Botulinum toxin injections within 3 months of research study
3. Medications with effects on the central nervous system including anticholinergic, benzodiazepines, and muscle relaxants among others within 1 week of the study
4. No physical or occupational therapy of the upper extremities
5. Any contraindications to MRI (ie: metal in body or implanted medical devices, etc)
6. Any contraindication on TMS adult safety screening (TASS form) including seizure history, pregnancy, brain injury, cranial metal implants, known structural brain lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of accurately delivering TMS during the task of writing as measured by number of participants who completed the TMS sessions | Visit 3 (week 1), Visit 4 (week 2), Visit 5 (week 3)

SECONDARY OUTCOMES:
Safety, as measured by TMS acute side effects | Visit 3 (week 1), Visit 4 (week 2), Visit 5 (week 3)
Feasibility, as measured by change in behavioral writing measure | Visit 3 (week 1), Visit 4 (week 2), Visit 5 (week 3)
  Using change in peak accelerations to assess writing behavior and further develop this writing behavior assessment tool throughout the study.
Change in brain connectivity in the motor network | Visit 3 (week 1), Visit 4 (week 2), Visit 5 (week 3)
  using functional magnetic resonance imaging of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Bukhari-Parlakturk, MD PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulcahey PJ, Peterchev AV, Calakos N, Bukhari-Parlakturk N. Transcranial magnetic stimulation: the road to clinical therapy for dystonia. Dystonia. 2023 August; 2.
- [Background] Bukhari-Parlakturk N, Mulcahey PJ, Lutz M, Ghazi R, Huang Z, Dannhauer M, Simsek Z, Groves S, Lipp M, Fei M, Tran T, Wood E, Beynel L, Scott B, Termsarasab P, Petty C, Al-Khalidi HR, Voyvodic J, Appelbaum LG, Davis S, Michael A, Peterchev AV, Calakos N. Functional MRI-guided personalized TMS decreases basal ganglia activity and improves focal hand dystonia. International Organization of Human Brain Mapping Conference. Montreal, Canada. July 22-26, 2023. virtual poster presentation.
- [Background] Bukhari-Parlakturk N, Mulcahey PJ, Lutz M, Ghazi R, Huang Z, Dannhauer M, Simsek Z, Groves S, Lipp M, Fei M, Tran T, Wood E, Beynel L, Scott B, Termsarasab P, Petty C, Al-Khalidi HR, Voyvodic J, Appelbaum LG, Davis S, Michael A, Peterchev AV, Calakos N. Functional MRI-guided personalized TMS decreases basal ganglia activity and improves focal hand dystonia. International Dystonia Symposium. Dublin, Ireland. June 1-3, 2023. poster presentation.
- [Background] Bukhari-Parlakturk N, Lutz MW, Al-Khalidi HR, Unnithan S, Wang JE, Scott B, Termsarasab P, Appelbaum LG, Calakos N. Suitability of Automated Writing Measures for Clinical Trial Outcome in Writer's Cramp. Mov Disord. 2023 Jan;38(1):123-132. doi: 10.1002/mds.29237. Epub 2022 Oct 13. PMID 36226903
- [Background] Dannhauer M, Huang Z, Beynel L, Wood E, Bukhari-Parlakturk N, Peterchev AV. TAP: targeting and analysis pipeline for optimization and verification of coil placement in transcranial magnetic stimulation. J Neural Eng. 2022 Apr 21;19(2):10.1088/1741-2552/ac63a4. doi: 10.1088/1741-2552/ac63a4. PMID 35377345